CLINICAL TRIAL: NCT07147946
Title: Evaluation of a Multicenter, Randomized, Double-Blind, Placebo-Controlled Phase III Clinical Trial on the Efficacy and Safety of Inhaled TQC3721 Suspension in Patients With Moderate-to-Severe Chronic Obstructive Pulmonary Disease
Brief Title: Evaluation of the Clinical Trial of Inhaled TQC3721 Suspension in Patients With Moderate-to-Severe Chronic Obstructive Pulmonary Disease
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TQC3721-III-01
Record Dates: First submitted 2025-08-22; First posted 2025-08-29 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-06

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Inhalation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TQC3721 Suspension for Inhalation (Experimental): Inhalation of TQC3721 suspension (6mg/2ml), one unit dose twice daily for 24 weeks
  Interventions: Drug: TQC3721 Suspension for inhalation
- Placebo of TQC3721 Suspension for Inhalation (Placebo Comparator): Inhalation of TQC3721 placebo, one unit dose twice daily for 24 weeks
  Interventions: Drug: Placebo of TQC3721 Suspension for Inhalation

INTERVENTIONS:
Drug: TQC3721 Suspension for inhalation — TQC3721 suspension for inhalation is a Phosphodiesterase3/4 (PDE3/4) inhibitor
  Arms: TQC3721 Suspension for Inhalation
Drug: Placebo of TQC3721 Suspension for Inhalation — Placebo without drug substance
  Arms: Placebo of TQC3721 Suspension for Inhalation

SUMMARY:
To evaluate the efficacy of TQC3721 Suspension for Inhalation in patients with moderate to severe Chronic obstructive pulmonary disease (COPD)

ELIGIBILITY:
Inclusion Criteria:

1. Sign an informed consent form before screening and fully understand the trial content, process, and potential adverse reactions.
2. Comply with the experimental schedule and be able to use the nebulizer inhaler correctly.
3. The age range is 40 to 80 years old (including the threshold), and both male and female participants are eligible.
4. The subjects have no pregnancy plans and voluntarily take effective contraceptive measures for at least one month from screening to the last use of the study drug.
5. Patients with a clear clinical history and related symptoms of COPD before screening.
6. Capable of conducting acceptable and reproducible lung function tests.
7. COPD clinical stability (no moderate to severe COPD acute exacerbation) within the 4 weeks prior to screening visit (V1 visit) and between V1 visit and V2 visit.
8. Smoking history ≥ 10 pack years.

Exclusion Criteria:

1. A history of life-threatening COPD, including admission to the intensive care unit and/or the need for intubation.
2. COPD acute exacerbations requiring systemic hormone therapy within 3 months prior to screening visit (V1 visit) or prior to randomization visit (V2 visit).
3. Within the first 6 months of screening, there has been at least 1 hospitalization history due to acute exacerbation of COPD or pneumonia.
4. Treatment with antibiotics for upper and/or lower respiratory tract infections within 6 weeks prior to screening or randomization visit (V3 visit).
5. Simultaneously suffering from other respiratory diseases.
6. Chest computed tomography (CT) revealed clinically significant abnormalities and concluded that the abnormalities were not caused by COPD.
7. Previous lung resection or lung reduction surgery.

11.Previously received TQC3721 treatment. 12.Patients who received immunosuppressant therapy within 4 weeks prior to the screening period 13.In the investigator's assessment, patients are unable to discontinue the prohibited drugs specified in the protocol during the screening and treatment phases of the study; 14.Patients with a history of uncontrolled current diseases that the investigator judges to be clinically significant; 15.A history or current evidence of clinically significant cardiovascular or cerebrovascular diseases; 16.A history of malignant tumors (cured or uncured) in any organ or system within the past 5 years; 17.Intolerance or allergy to salbutamol or other inhaled bronchodilator therapies for COPD; 18.Patients requiring long-term oxygen therapy; 19.Female subjects who are currently pregnant, breastfeeding, or planning to become pregnant during the study period after enrollment; 20.Having participated in any clinical trial of drugs or medical devices within 4 weeks or 5 half-lives (whichever is longer) prior to the screening visit; 21.Other conditions deemed unsuitable for participation in the study by the investigator.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 666 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Mean change in the area under the curve (AUC) of Forced Expiratory Volume in 1 second (FEV1) | Baseline to 12 weeks after treatment
  Change from baseline in mean FEV1 AUC over 0-12 hours after 12 weeks of treatment.

SECONDARY OUTCOMES:
Changes in peak FEV1 value | Baseline to 6 weeks, 12 weeks, 24 weeks after treatment
  Changes from baseline in peak FEV1 within 4 hours after morning dosing at Weeks 6, 12, and 24 of treatment.
Changes in trough FEV1 values | Baseline to 6 weeks, 12 weeks, 24 weeks after treatment
  Changes from baseline in morning trough FEV1 at Weeks 6, 12, and 24 of treatment.
Average FEV1 AUC 0-4h | Baseline to 6 weeks, 12 weeks, 24 weeks after treatment
  Change from baseline in the average FEV1 AUC 0-4h within 4 hours after morning dosing at 6, 12, and 24 weeks of treatment.
St. George's Respiratory Questionnaire | Baseline to 6 weeks, 12 weeks, 24 weeks after treatment
  Changes in St. George's Respiratory Questionnaire (SGRQ) total scores from baseline at 6, 12, and 24 weeks of treatment.
Chronic Obstructive Pulmonary Disease Assessment Test | At 6 weeks, 12 weeks, and 24 weeks of treatment
  Self-assessment for Patients with COPD：Numbers 0 to 5 indicate the severity (with 0 being the mildest and 5 being the most severe).
Average FEV1 AUC (6-12h) | Baseline to 12 weeks after treatment
  Change from baseline in mean FEV₁ AUC (6-12 h) at Week 12 following dosing.
Annual rate of acute exacerbation of COPD | Baseline to 24 weeks after treatment
  The annualized rate of acute exacerbation of moderate/severe COPD after 24 weeks of treatment.
Time of first acute exacerbation of moderate/severe COPD | Baseline to 24 weeks after treatment
  The time of the first acute exacerbation of moderate/severe COPD within 24 weeks of treatment.
Adverse event (AE) | D-28 to within 25 weeks of treatment
  The number of participants with AEs, serious dverse event (SAEs), drug-related AEs, and abnormal lab results.
Assessment of respiratory symptoms in COPD | Baseline to 6 weeks, 12 weeks, 24 weeks after treatment
  Change from baseline in weekly mean Evaluating Respiratory Symptoms in COPD total score
Transition Dyspnea Index (TDI) score | Baseline to 6 weeks, 12 weeks, 24 weeks after treatment
  Change in Transition Dyspnea Index (TDI) score relative to Baseline Dyspnea Index (BDI) score
Chronic Obstructive Pulmonary Disease Assessment Test (CAT) score | Baseline to 6 weeks, 12 weeks, 24 weeks after treatment
  Change in Chronic Obstructive Pulmonary Disease Assessment Test (CAT) score from baseline
Change from baseline in rescue medication use | Baseline to 6 weeks, 12 weeks, 24 weeks after treatment.
  Changes from baseline in rescue medication use during treatment at Weeks 6, 12, and 24 versus the placebo group
Interleukin-6 (IL-6), Interleukin-8 (IL-8), and C-reactive protein (CRP) at Week 12 and Week 24 | At Week 12 and Week 24
  IL-6, IL-8, and C-reactive protein (CRP) at Week 12 and Week 24. The elevated serum C-reactive protein (CRP) levels in patients with chronic obstructive pulmonary disease (COPD) are primarily associated with pulmonary inflammatory responses.
Plasma drug peak concentration | Day 1: 0.5 hour after-dose, Week 6: 1 hour pre-dose, 0.5 hour after-dose; Week 12: 1 hour pre-dose, 0.5 hour after-dose
  Perform Pharmacokinetics (PK) analysis of TQC3721 blood drug concentration data at baseline, week 6, and week 12 to evaluate the PK characteristics of TQC3721 in COPD patients.

CONTACTS AND LOCATIONS:
Locations (76):
- China (76):
  - Bozhou People's Hospital, Bozhou, Anhui
  - Chizhou People's Hospital, Chizhou, Anhui
  - Chaohu Hospital of Anhui Medical University, Hefei, Anhui
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Peolpe's Hospital Of Chongqing Banan District, Chongqing, Chongqing Municipality
  - Chongqing University Three Gorges Hospital, Chongqing, Chongqing Municipality
  - Fuling Hospital Affiliated to Chongqing University, Chongqing, Chongqing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Zhangzhou Municipal Hospital of Fujian Province, Zhangzhou, Fujian
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - Gansu Provincial Hospital, Lanzhou, Gansu
  - The Eighth Affiliated Hospital of Southern Medical University（The First people's Hospital of Shunde ）, Foshan, Guangdong
  - Huizhou Central People's Hospital, Huizhou, Guangdong
  - Longgang District People's Hospital of Shenzhen, Shenzhen, Guangdong
  - Peking University Shenzhen Hospital, Shenzhen, Guangdong
  - Guizhou Provincial People's Hospital, Guiyang, Guizhou
  - The First Affiliated Hospital of Hainan Medical University, Haikou, Hainan
  - Cangzhou Hospital of Integrated TCM- WM·HEBEI, Cangzhou, Hebei
  - Hebei PetroChina Central Hospital, Langfang, Hebei
  - The First Hospital of Qinhuangdao, Qinhuangdao, Hebei
  - Hebei Medical University Third Hospital, Shijiazhuang, Hebei
  - Daqing Longnan Hospital, Daqing, Heilongjiang
  - The First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Qiqihar First Hospital, Qiqihar, Heilongjiang
  - Jiaozuo Second People's Hospital, Jiaozuo, Henan
  - Puyang Oilfield General Hospital, Puyang, Henan
  - The First People's Hospital of Shangqiu, Shangqiu, Henan
  - Yichang Central People's Hospital, Yichang, Hubei
  - Hunan Provincial People's Hospital, Changsha, Hunan
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - The Central Hospital of Yongzhou, Yongzhou, Hunan
  - Baotou Central Hospital, Baotou, Inner Mongolia
  - Chifeng Municipal Hospital, Chifeng, Inner Mongolia
  - Inner Mongolia Medical University Affiliated Hospital, Hohhot, Inner Mongolia
  - Nanjing Jiangning Hospital, Nanjing, Jiangsu
  - The Fifth People's Hospital of Wuxi, Wuxi, Jiangsu
  - Jiangyin Hospital of Traditional Chinese Medicine, Wuxi, Jiangsu
  - Xuzhou Central Hospital, Xuzhou, Jiangsu
  - Subei People's Hospital of Jiangsu province, Yangzhou, Jiangsu
  - Yixing People's Hospital, Yixing, Jiangsu
  - Jiujiang First People's Hospital, Jiujiang, Jiangxi
  - Jiangxi Provincial People's Hospital, Nanchang, Jiangxi
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The first hospital of Jilin University, Changchun, Jilin
  - Central Hospital of Dalian University of Technology, Dalian, Liaoning
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Qinghai Provincial People's Hospital, Xining, Qinghai
  - Xi'an International Medical Center Hospital, Xi'an, Shaanxi
  - Yan'an University Xianyang Hospital, Xianyang, Shaanxi
  - Binzhou People's Hospital, Binzhou, Shandong
  - Heze Municipal Hospital, Heze, Shandong
  - Affiliated Hospital of Jining Medical University, Jining, Shandong
  - Weifang NO.2 People's Hospital, Weifang, Shandong
  - Yantai Yuhuangding Hospital, Yantai, Shandong
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai General Hospital, Shanghai, Shanghai Municipality
  - Baoji Central Hospital, Baoji, Shanxi
  - Changzhi People's Hospital, Changzhi, Shanxi
  - Yangquan coal Industry(Group) General Hospital, Yangquan, Shanxi
  - The First Affiliated Hospital of Chengdu Medical College, Chengdu, Sichuan
  - Chengdu Second People's Hospital, Chengdu, Sichuan
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Mianyang Central Hospital, Mianyang, Sichuan
  - Mianyang Hospital of Traditional Chinese Medicine, Mianyang, Sichuan
  - Affiliated Hospital of North Sichuan Medical College, Nanchong, Sichuan
  - Suining Central Hospital, Suining, Sichuan
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - Tianjin 4th Center Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Shihezi University, Shihezi, Xinjiang
  - The Second Hospital of Jiaxing, Jiaxing, Zhejiang
  - Jinhua municipal central hospital, Jinhua, Zhejiang
  - Dongyang People's Hospital, Jinhua, Zhejiang
  - The First Affiliated Hospital of Ningbo University, Ningbo, Zhejiang
  - Shaoxing People's Hospital, Shaoxing, Zhejiang
  - Taizhou Central Hospital, Taizhou, Zhejiang
  - The Second Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang